CLINICAL TRIAL: NCT02008981
Title: A Randomized, Double Blind, Placebo-controlled Crossover Study on the Effect of Commonly Used Herbal Products on Platelet Function and Coagulation Profile of Healthy Volunteers
Brief Title: Effect of Herbal Products on Platelet Function and Clotting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM platelet function
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Platelet Function Test
MeSH Terms: interventions — turmeric extract; angelicae sinensis extract; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Angelica sinensis (Active Comparator): Angelica sinensis in capsule form will be given with actual or placebo aspirin, each for a 3 week period. Clotting profile and platelet function test will be done before and after.
  Interventions: Drug: Angelica sinensis; Drug: Aspirin
- Curcuma longa (Active Comparator): Curcuma longa in capsule form will be given with actual or placebo aspirin, each for a 3 week period. Clotting profile and platelet function test will be done before and after.
  Interventions: Drug: Curcuma longa; Drug: Aspirin
- Siwu Tang (Active Comparator): TCM formulation "Siwu Tang" consisting of 4 herbs ( Ligustici chuangxiong, Angelicae sinensis, Rehmanniae praeparata and Paeoniae alba) in tablet form will be given with actual or placebo aspirin, each for a 3 week period. Clotting profile and platelet function test will be done before and after.
  Interventions: Drug: Siwu Tang; Drug: Aspirin

INTERVENTIONS:
Drug: Curcuma longa — Curcuma longa in capsule form will be given with actual or placebo aspirin, each for a 3 week period. Clotting profile and platelet function test will be done before and after.
  Arms: Curcuma longa
Drug: Angelica sinensis — Angelicae sinensis in capsule form will be given with actual or placebo aspirin, each for a 3 week period. Clotting profile and platelet function test will be done before and after.
  Arms: Angelica sinensis
Drug: Siwu Tang — TCM formulation "Siwu Tang" consisting of 4 herbs ( Ligustici chuangxiong, Angelicae sinensis, Rehmanniae praeparata and Paeoniae alba) in tablet form will be given with actual or placebo aspirin, each for a 3 week period. Clotting profile and platelet function test will be done before and after.
  Arms: Siwu Tang
Drug: Aspirin — Aspirin (enteric-coated) at 100mg daily will be given one of the actual herb or placebo herb, each for a 3 week period. Clotting profile and platelet function test will be done before and after.

SUMMARY:
This is a research study on the effect of some commonly used "blood activating" herbal products on platelet function and coagulation profile, ie whether it causes an increase in bleeding tendency, either used alone or in combination with Aspirin which is a commonly used anti-platelet drug.

DETAILED DESCRIPTION:
This study is being conducted because there has not been any proper studies to provide evidence that these commonly used "blood activating" herbal preparations can in fact affect blood clotting by interfering with platelet function or clotting mechanism and potentiate the antiplatelet activity of Aspirin. These are assumptions based on TCM theory, laboratory experiments and animal studies but have led to the general statement in medical literature that these herbs increases bleeding risk in patients taking Aspirin or any other anti-platelet drugs. This has resulted in advice that these herbal products should not be taken by patients on Aspirin, which is a common drug taken by many patients. We hope to prove or disprove this theoretical concern by measurement of platelet and clotting function in healthy volunteers before and after taking the herbal product, alone and in combination with Aspirin. This will help to answer the question of whether it is safe for patients to take these common "blood -activating " herbs alone or together with Aspirin.

Healthy volunteers will be consecutively enrolled into 3 arms, each studying one herbal product for 25 volunteers. The design involves taking all 3 of the following combinations: aspirin + placebo, herb + placebo, aspirin + herb, each for a 3-week period, in a randomized order, with 2 weeks of wash-out in between each 3-week period. Platelet function and coagulation profile will be assayed

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18 and 70 years.
2. Healthy by medical history and physical exam.
3. Laboratory values within established guidelines for participation in clinical studies: AST less than or equal to 2 times the ULN; SCr less than or equal to ULN; FBC showing normal Hb; WBC and platelet count; normal aPTT/PT
4. Negative urine pregnancy test for females of child-bearing potential.
5. Females of child-bearing potential who are able and willing to practice abstinence or use non-hormonal effective methods of birth control during the study, such as condoms or diaphragms.

Exclusion Criteria:

1. Concomitant therapy (chronic or intermittent) with herbal drugs, aspirin, any other anti-platelet agents, non-steroidal anti-inflammatory medications or warfarin from 14 days prior to study participation and throughout the study period
2. Inability to obtain venous access for blood sample collection.
3. The presence of any of the following significant medical conditions:

   1. Diabetes mellitus poorly controlled or requiring insulin
   2. Hypertension poorly controlled
   3. Cardiac disease : heart failure, arrhythmia poorly controlled
   4. Renal disease,
   5. Hepatic impairment
   6. Bleeding disorders including thrombocytopenia and coagulopathy, either congenital or acquired
   7. Peptic ulcer disease
   8. Psychiatric illnesses that may interfere with the subject's ability to participate in the study, or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigators.
4. Plans for elective surgery during the investigation or within 2 weeks following completion of the study.
5. Positive urine pregnancy test or breastfeeding female.
6. The presence of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.
7. Drug or alcohol abuse that may impair safety or adherence (more than 3 alcoholic drinks per day, on a daily basis).
8. History of intolerance or allergic reaction to aspirin or any NSAIDS
9. Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
platelet function test and coagulation profile | 3 weeks
  Platelet function test and coagulation profile ( aPTT/PT) will be done at baseline and after each phase of 3 weeks of Herb/aspirin or their placebo

CONTACTS AND LOCATIONS:
Overall Officials: Yeh-Ching Linn, MBBS, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore